CLINICAL TRIAL: NCT07210372
Title: Post-Operative Axial Stabilty in Short and Long Eyes After Implanation of a Clareon Intraocular Lens
Brief Title: Axial Stability in Short and Long Eyes After Cataract Surgery
Acronym: ACDC
Status: Completed | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: JKU-Ophthalmology-002-ACDC
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Introcular Lens Position
Keywords: intraocular lens position; lens position; axial length; short eye; long eye; cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- short eye: patients with eye length up to 22,75mm
- long eye: patients with eye length at least 25,50mm

SUMMARY:
Post operative intraocular lens position is being measured after cataract surgery in 34 patients with long and short eyes.

DETAILED DESCRIPTION:
Prediction of the post-operative IOL position in long and short eyes the prediction difficult. Therefore, it is relevant to evaluate the post-operative IOL position in patients with an axial eye length outside the typical range. This study will help to improve the prediction of the post-operative refractive outcome in short and long eyes after implantation of a Clareon IOL. Therefore, three different OCT based measurements will be used (IOLMaster700, CZM; CASIA II, Tomey; SM-39, CSO), respectively. Post-operatively, these measurements will be repeated 1 hour, 1 week, and 12 weeks after surgery.

Hypothesis: Implantation of the Clareon IOL leads to a stable post-operative IOL position in short (≤22.75mm) and long (≥25.50mm) eyes.

Endpoints:

Primary Endpoint: change in anterior chamber depth (=IOL position) in mm from 1 week to 12 weeks post-operative visit for both short and long eyes (two separate analysis) (Refraction will be a secondary outcome due to its larger variability compared to ACD measurements 1)

Secondary Endpoint:

* Refractive outcome after Clareon IOL implantation at 1- and 12-week visit o
* Monocular BCDVA and DCIVA (66cm) at 1 week and 12-week post-operative visit

  o Subjects with a post operative tilt (at 12-week post operative visit) ≥10⁰ will be excluded from VA analysis
* Change in ACD in mm from 1 hour to 12 weeks, 1 hour to 1-week post-op visit for both short and long eyes Exploratory Endpoints
* Comparison of refractive outcome between long and short eyes via prediction error for Barret Universal II for long eyes and Kane formula for short eyes with target emmetropia to -2.50D based on subject's visual needs ACD in mm 1 hour, 1 week, and 12 weeks post op as measured from corneal epithelium to anterior lens surface by IOL master 700, Casia II, and MS 39

Principal Objective: Aim of this study is to measure the change in the post-operative Anterior Chamber Depth of the Clareon monofocal IOL in short/long eyed patients at different post operative time points (1 hour, 1 week, and 12 weeks) during uneventful FLACS cataract surgery.

* Exploratory/secondary Objectives:
* To measure post-operative monocular corrected visual acuity of the Clareon IOL at distance and intermediate vision (66cm)
* To Compare refractive outcomes between long and short eyes

ELIGIBILITY:
Inclusion Criteria:

* bilateral cataract surger
* axial eye length below 22,75mm or above 25.50mm

Exclusion Criteria:

* ocular pathologies that could lead to an unstable capsular bag
* pregnancy
* preoperative visual acuity above 1.0logMar

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients undergoing planned cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
change in anterior chamber depth | 1 week and 12 weeks post operative
  change in anterior chamber depth in millimeter

SECONDARY OUTCOMES:
refractive outcome after intraocular lens implantation | 1 week and 12 weeks post operative
  spherical equivalent

CONTACTS AND LOCATIONS:
Overall Officials: Nino Hirnschall, MD, Principal Investigator — Kepler Universitätsklinikum /JKU
Locations (1):
- Kepler University Clinic, Linz, Linz, Austria